CLINICAL TRIAL: NCT01284790
Title: Pitch and Loudness Perception by Cochlear Implant Listeners: Psychophysics and Objective Measures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-A00439-30; 2009-35 (Other: AP HM)
Record Dates: First submitted 2011-01-21; First posted 2011-01-27 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Cochlear Implant Listeners
MeSH Terms: interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cochlear implants (Experimental)
  Interventions: Device: Cochlear implants

INTERVENTIONS:
Device: Cochlear implants

SUMMARY:
Cochlear implants (CIs) have restored some sense of hearing to more than 120 000 people worldwide. While most patients show good scores of speech recognition in quiet, a large majority of them also struggle in more challenging listening situations, such as speech in noise or music. This project aims to understand the basic mechanisms of electrical stimulation of the auditory nerve, in order to identify the important cues that the electrical signal should convey and to possible improve sound perception by CI users.

DETAILED DESCRIPTION:
This study will take place in the ENT department of La Timone hospital in Marseille, where more than 120 adults have been implanted. Our study will comprise several phases, including (1) temporal coding of pitch, (2) spatial coding of pitch, and (3) loudness perception. Eight adult implant users will be recruited for each of these phases.

ELIGIBILITY:
Inclusion Criteria:

* The adults of more than 18 years old at the beginning of the study without notion of minimal or maximal duration of setting-up(presence).
* The adults WITH cochlear implant listeners .

Exclusion Criteria:

* Presence of intrusive disorders of the personality or mental deficiency. Presence of associated driving disorders. Pregnant or breast-feeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Identify waveforms aimed to improve sound perception by CI recipients | 2 YEARS

SECONDARY OUTCOMES:
To correlate the results of our measures psychophysiques with recordings électrophysiologiques of the neuronal activity of the hearing nerve. | 2 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France